CLINICAL TRIAL: NCT05059626
Title: Mechanisms and Interventions Addressing Accelerated Cardiovascular Disease Risk in Women With Endometriosis
Brief Title: Endometriosis and Microvascular Dysfunction; Simvastatin and Duavee
Acronym: Endo2/SA3
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: The John B. Pierce Laboratory (Other)
Responsible Party: Principal Investigator, Lacy Alexander, Professor of Kinesiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18347
Record Dates: First submitted 2021-09-10; First posted 2021-09-28 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis
Keywords: Skin blood flow; Estrogen; Selective Estrogen Receptor Modulator; Intradermal Microdialysis
MeSH Terms: conditions — Endometriosis | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: This is a single arm randomized study. Only women with endometriosis will complete this study. Once consented and screened, each subject is block randomized to either 30 days of a treatment (Simvastatin or 30 days of SERM (bazedoxifene + conjugated estrogen; BZE+CE)). This will be done in a counterbalanced fashion. Subjects will have the option of completing the other arm of the study but will undergo a 60 day washout to mimimize carry over effect. We will use Research Randomizer software. These treatments are blinded to the investigators collecting the data and performing the data analysis.
Who Masked: Investigator
Masking Description: These treatments are blinded to the investigators. The subjects, physician, and the nurse on staff knows which treatment the subject is taking if there are any questions or safety concerns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Simvastatin (Other): 30 days of Simvastatin (10mg/day)
  Interventions: Drug: simvastatin 10mg
- bazedoxifene + conjugated estrogen (Other): 30 days of bazedoxifene + conjugated estrogen (0.45mg/20mg/day)
  Interventions: Drug: Bazedoxifene 20/Estrogens,Con 0.45Mg Tb

INTERVENTIONS:
Drug: simvastatin 10mg — Simvastation acts as a systemic LOX inhibitor.
  Arms: Simvastatin
Drug: Bazedoxifene 20/Estrogens,Con 0.45Mg Tb — Duavee is a selective estrogen receptor modulator.
  Arms: bazedoxifene + conjugated estrogen

SUMMARY:
Purpose: To determine the effects of SERM and simvastatin interventions on endothelial dysfunction in women with endometriosis.

Hypothesis: Treatment with the SERM (bazedoxifene + conjugated estrogen) or with simvastatin will decrease systemic inflammation and improve specific measures of cardiovascular function including endothelium-dependent vasodilation.

DETAILED DESCRIPTION:
Endometriosis is an estrogen dependent gynecological disorder associated with considerable chronic pelvic pain, pain during intercourse and is a major cause of infertility. While endometriosis is a local inflammatory syndrome, the inflammatory process is systemic and underlies many of the co-morbidities associated with this devastating disease. Endometriosis and atherosclerotic cardiovascular disease (CVD) are both inflammation-induced diseases. Robust epidemiologic data demonstrate a clear association between endometriosis, reproductive risk factors, inflammation and CVD risk, the leading cause of death in women worldwide. Estrogen exposure is beneficial for women from a CVD standpoint, but the standard of treatment for endometriosis includes estrogen suppression. This creates a conundrum for the long-term management of CVD risk in women with endometriosis. Moreover, there is a significant gap in prior research into the role of inflammatory signaling, CVD risk and effective interventions to mitigate cardiovascular comorbidities.

Endometriosis and Endothelial Dysfunction: Circulating LDL and oxidized (ox)LDL are two of many biomarkers of cardiovascular and inflammatory disease elevated in women with endometriosis. These circulating factors and inflammatory cytokines stimulate the ubiquitously expressed scavenger lectin-like oxidized LDL receptor (LOX-1) on the vasculature resulting in increased oxidant production and reduced nitric oxide (NO) metabolism, resulting in pronounced endothelial dysfunction, one of the earliest detectable indicators of increased CVD risk. Interestingly, estrogen directly inhibits LOX-1-dependent endothelial dysfunction. Our working model is that endometriosis-associated systemic inflammatory mediators increase LOX-1 receptor activity and result in endothelial dysfunction.

Therapies approved in 2018 for the treatment of endometriosis reduce endogenous estrogen production (elagolix) or selectively modulate estrogen receptors (SERM, bazedoxifene). Additionally, in preclinical models, therapies that modulate vascular function (statins) are also efficacious for reducing endometriosis proliferation. However, to date no studies have evaluated outcomes specific to systemic inflammation and cardiovascular function with these emerging endometriosis therapies.

This is a single arm pre/post study design. Only women with endometriosis will complete this study. Women will be between the ages of 18 and 45 years and previously diagnosed (within the past 5 years) with endometriosis. Once consented and screened, each subject is block randomized to either 30 days of a treatment (Simvastatin or 30 days of SERM (bazedoxifene + conjugated estrogen; BZE+CE)) and , or statin. This will be done in a counterbalanced fashion. Subjects will only complete one of the treatments and the placebo with a 60 day washout to minimize potential carryover effects. On day 30 of pretreatment , each subject participates in a cutaneous microdialysis (MD) and flow mediated dilation (FMD) experiment. After a 60-day washout, the participant will start either the treatment or placebo and returns to repeat the study with the other pre-treatments (SERM/Statin/Placebo)undergo the MD and FMD experiments. These treatments/placebo are blinded to the investigators collecting and analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 45 years with endometriosis (diagnosis by prior laparoscopy by subject's own physician <10 years prior, and reported by the subject to the researchers)
* Tylenol if the subject has acute pain is allowed
* IUD contraceptive use (copper or levonogestrel) is allowed

Exclusion Criteria:

* Use of nicotine-containing products (e.g. smoking, chewing tobacco, etc.)
* Diabetes (HbA1C .6.5%)
* BP>140/90
* Taking pharmacotherapy that could alter peripheral vascular control (e.g. insulin sensitizing, cardiovascular medications)
* Pregnancy
* Breastfeeding
* Taking illicit and/or recreational drugs
* Abnormal liver function
* Rash, skin disease, disorders of pigmentation, known skin allergies
* Diagnosed or suspected metabolic or cardiovascular disease
* Persistent unexplained elevations of serum transaminases
* Known allergy to latex or investigative substances

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in skin blood flow | before intervention and 30 days post-intervention
  cutaneous vascular conductance (units = red cell flux/mean arterial pressure)
Change in peripheral blood flow | before intervention and 30 days post-intervention
  brachial artery flow mediated dilation

SECONDARY OUTCOMES:
Change in LOX-1 activity | before intervention and 30 days post-intervention
  LOX-1 receptor expression
Change in reproductive hormones | before intervention and 30 days post-intervention
  blood hormone concentrations
Change in inflammation | before intervention and 30 days post-intervention
  inflammatory cytokine concentration
Change in microRNA activity | before intervention and 30 days post-intervention
  microRNA expression

CONTACTS AND LOCATIONS:
Locations (1):
- The John B. Pierce Laboratory, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No